CLINICAL TRIAL: NCT00121836
Title: An Open-label Study of Xeloda Plus Avastin at Time of Disease Progression in Treatment-naïve Women With HER2-negative Metastatic Breast Cancer
Brief Title: A Study of Xeloda (Capecitabine) in Women With HER2-Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Disclosures Group, Hoffmann-La Roche
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18527
Record Dates: First submitted 2005-07-18; First posted 2005-07-21 (Estimated); Results first posted 2011-03-04 (Estimated); Last update posted 2011-04-27 (Estimated); Status verified 2011-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Bevacizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Capecitabine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Capecitabine — 1000 mg/m² PO BID on Days 1-15 of each 3-week cycle
  Other Names: Xeloda
Drug: Bevacizumab — 15 mg IV on Day 1 of each 3-week cycle
  Other Names: Avastin

SUMMARY:
This single-arm study was designed to evaluate the efficacy and safety of oral Xeloda plus intravenous Avastin as first-line treatment in women with metastatic breast cancer. Patients received Xeloda 1000 mg/m² orally (PO) twice daily (BID) on Days 1-15, and Avastin 15 mg intravenously (IV) on Day 1 of each 3-week cycle. The anticipated time on study treatment was until disease progression or unacceptable toxicity. The target sample size was <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* Women >=18 years of age
* HER2-negative metastatic breast cancer
* Previous adjuvant chemotherapy or hormonal treatment
* >=1 measurable target lesion

Exclusion Criteria:

* Previous treatment with chemotherapy, an anti-angiogenic agent, or a biologic therapy for advanced or metastatic cancer
* Radiation therapy within 4 weeks of study treatment start or insufficient recovery from the effects of prior radiation therapy
* Central nervous system metastases
* Other malignancy within last 5 years, except cured basal cell carcinoma of skin and carcinoma in situ of uterine cervix
* Serious concurrent infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2005-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (42):
- United States (42):
  - Birmingham, Alabama
  - Burbank, California
  - Glendale, California
  - Los Angeles, California
  - San Diego, California
  - Farmington, Connecticut
  - Bonita Springs, Florida
  - Boynton Beach, Florida
  - Bradenton, Florida
  - Cape Coral, Florida
  - Fort Myers, Florida
  - Naples, Florida
  - Port Charlotte, Florida
  - Sarasota, Florida
  - Venice, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Tucker, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Waterloo, Iowa
  - Scarborough, Maine
  - Prince Frederick, Maryland
  - Lansing, Michigan
  - Kansas City, Missouri
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Brick, New Jersey
  - Neptune City, New Jersey
  - Red Bank, New Jersey
  - Rochester, New York
  - Hickory, North Carolina
  - Canton, Ohio
  - Oklahoma City, Oklahoma
  - Beaufort, South Carolina
  - Charleston, South Carolina
  - Florence, South Carolina
  - Hilton Head Island, South Carolina
  - Sumter, South Carolina
  - Abingdon, Virginia
  - Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Capecitabine+Bevacizumab (Bev); Paclitaxel or Vinorelbine +Bev: First Study Treatment Phase:
  Capecitabine 1000 mg/m² oral (PO) twice-daily, Days 1-15 of each 3-week cycle (28 doses per cycle); bevacizumab 15 mg/kg intravenous (IV) infusion, Day 1 of each 3-week cycle.
  Second Study Treatment Phase:
  Paclitaxel 80 mg/m² 60-minute IV infusion (with appropriate premedication), Days 1, 8 and 15 of each 4-week cycle (28 days). Substitution of paclitaxel with docetaxel was not allowed.
  Vinorelbine 25 mg/m² IV infusion over 10-20 minutes, Days 1, 8, and 15 of each 4-week cycle.
  Bevacizumab 10 mg/kg IV infusion, Days 1 and 15 of each 4-week cycle.
Period: Overall Study
Arm/Group | Capecitabine+Bevacizumab (Bev); Paclitaxel or Vinorelbine +Bev
Started | 109
Completed | 54
Not Completed | 55

BASELINE CHARACTERISTICS:
Arm/Group | Capecitabine+Bevacizumab (Bev); Paclitaxel or Vinorelbine +Bev
Number analyzed (Participants) | 109
Age Continuous [Mean (Standard Deviation); unit: Years] | 56.7 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time from date of first treatment dose (Day 1) to date of death, across the study phases regardless of the cause of death
Time Frame: approximately 505 days (Median Time to Death)
Population: 109 patients (pts) received study drug in the First Study Treatment Phase. 54 pts withdrew prematurely, and 54 pts proceeded to the Second Study Treatment Phase. All 54 pts who proceeded to the Second Study Treatment Phase withdrew during that phase. 1 pt continued treatment in the First Study Treatment Phase and completed 3 years of follow-up.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Capecitabine+Bevacizumab (Bev); Paclitaxel or Vinorelbine +Bev
Number analyzed (Participants) | 109
Days | 505 [420 to 672]

2. Secondary Outcome: Number of Subjects With Adverse Events
Description: The secondary outcome measure was to evaluate the safety profile, including a summary of adverse events (AEs) assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0.
  Intensity of AEs were graded according to NCI CTCAE version 3.0 on a 5-point scale: Grade 1=Mild Discomfort, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life Threatening/Disabling and Grade 5=Death. An SAE was defined as any experience that suggested a significant hazard,contraindication, side effect, or precaution.
Time Frame: Throughout study
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- First Study Treatment Phase Only: Capecitabine+Bevacizumab:
  Capecitabine 1000 mg/m² oral (PO) twice-daily, Days 1-15 of each 3-week cycle (28 doses per cycle); bevacizumab 15 mg/kg intravenous (IV) infusion, Day 1 of each 3-week cycle.
Arm/Group | Capecitabine+Bevacizumab (Bev); Paclitaxel or Vinorelbine +Bev | First Study Treatment Phase Only
Number analyzed (Participants) | 109 | 55
Participants
  At least 1 adverse event (AE) | 108 | 54
  At least 1 treatment-related AE | 104 | 51
  At least 1 Grade 3 or 4 AE | 82 | 41
  At least 1 serious adverse event (SAE) | 39 | 22
  At least 1 AE causing withdrawal | 37 | 25

3. Secondary Outcome: Premature Withdrawal From Study Due to Adverse Events
Description: The secondary outcome measure was to evaluate the safety profile, including a summary of premature withdrawals due to adverse events occurring in more than 1 patient in either study group, by system organ class.
Time Frame: Throughout study
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Capecitabine+Bevacizumab (Bev); Paclitaxel or Vinorelbine +Bev | First Study Treatment Phase Only
Number analyzed (Participants) | 109 | 55
Participants
  All system organ classes | 25 | 37
  General disorders, administration site conditions | 4 | 7
  Musculoskeletal and connective tissue disorders | 2 | 6
  Respiratory, thoracic and mediastinal disorders | 2 | 5
  Renal and urinary disorders | 2 | 2

4. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities
Description: The secondary outcome measure was to evaluate the safety profile, including a summary of marked laboratory abnormalities in >= 5% of patients. n=number of participants with the laboratory measure,Number=number of participants with the abnormality. Laboratory values were flagged as Low(L) or High(H) if they were below the lower limit or above the upper limit of Roche standard reference range, respectively. Marked laboratory abnormalities (flagged as HH and LL) were defined as those values that were outside the Roche marked reference range and showed a clinically relevant change from baseline.
Time Frame: until progressive disease or for up to 3 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Capecitabine+Bevacizumab (Bev); Paclitaxel or Vinorelbine +Bev
Number analyzed (Participants) | 109
Participants
  Hematocrit (fraction) (n=104); Abnormality: Low | 16
  Hemoglobin (g/L) (n=104); Abnormality: Low | 18
  Platelets (10^9/L) (n=104); Abnormality: Low | 9
  Red blood cells (10¹²/L) (n=104); Abnormality: Low | 15
  White blood cells (10^9/L)(n=104); Abnormality:Low | 23
  Neutrophils (10^9/L) (n=92); Abnormality: High | 14
  Neutrophils (10^9/L) (n=92); Abnormality: Low | 25
  Prothrombin time (ratio) (n=36); Abnormality: High | 3
  Aspartate transaminase(U/L)(n=104)Abnormality:High | 19
  Alanine transaminase(U/L)(n=104);Abnormality: High | 10
  Alkaline phosphatase(U/L)(n=104);Abnormality: High | 11
  Direct bilirubin (umol/L) (n=78);Abnormality: High | 4
  Albumin (g/L) (n=104); Abnormality: Low | 13
  Total protein (g/L) (n=104); Abnormality: Low | 8
  Chloride (mmol/L) (n=104); Abnormality: Low | 5
  Calcium (mmol/L) (n=104); Abnormality: Low | 10
  Uric acid (umol/L) (n=94); Abnormality: High | 5

ADVERSE EVENTS:
Arm/Group | Capecitabine+Bevacizumab (Bev); Paclitaxel or Vinorelbine +Bev
Serious Adverse Events (participants affected / at risk) | 39/109
Other Adverse Events (participants affected / at risk) | 103/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine+Bevacizumab (Bev); Paclitaxel or Vinorelbine +Bev (N=109)
Pain (General disorders) | 6
Chest Pain (General disorders) | 3
Mucosal Inflammation (General disorders) | 2
Fatigue (General disorders) | 1
Influenza Like Illness (General disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Abdominal Pain (Gastrointestinal disorders) | 1
Caecitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Enterovesical Fistula (Gastrointestinal disorders) | 1
Gastric Ulcer (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Bacterial Sepsis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Perirectal Abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Decreased Appetite (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hip Fracture (Injury, poisoning and procedural complications) | 1
Scapula Fracture (Injury, poisoning and procedural complications) | 1
Cerebral Haemorrhage (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Blood Sodium Decreased (Investigations) | 1
Haemoglobin Decreased (Investigations) | 1
Urine Output Decreased (Investigations) | 1
Haemorrhage (Vascular disorders) | 1
Phlebitis (Vascular disorders) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Left Ventricular Failure (Cardiac disorders) | 1
Metastases to Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal Failure (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine+Bevacizumab (Bev); Paclitaxel or Vinorelbine +Bev (N=109)
Diarrhoea (Gastrointestinal disorders) | 66
Nausea (Gastrointestinal disorders) | 66
Constipation (Gastrointestinal disorders) | 41
Vomiting (Gastrointestinal disorders) | 36
Dyspepsia (Gastrointestinal disorders) | 25
Stomatitis (Gastrointestinal disorders) | 15
Abdominal Pain (Gastrointestinal disorders) | 12
Abdominal Pain Upper (Gastrointestinal disorders) | 8
Abdominal Distension (Gastrointestinal disorders) | 7
Oral Pain (Gastrointestinal disorders) | 6
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 71
Alopecia (Skin and subcutaneous tissue disorders) | 32
Rash (Skin and subcutaneous tissue disorders) | 21
Nail Disorder (Skin and subcutaneous tissue disorders) | 13
Pruritus (Skin and subcutaneous tissue disorders) | 12
Erythema (Skin and subcutaneous tissue disorders) | 10
Dry Skin (Skin and subcutaneous tissue disorders) | 9
Skin Reaction (Skin and subcutaneous tissue disorders) | 9
Fatigue (General disorders) | 68
Mucosal Inflammation (General disorders) | 30
Pyrexia (General disorders) | 21
Pain (General disorders) | 19
Asthenia (General disorders) | 13
Oedema Peripheral (General disorders) | 13
Chills (General disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 29
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 28
Back Pain (Musculoskeletal and connective tissue disorders) | 21
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 17
Bone Pain (Musculoskeletal and connective tissue disorders) | 9
Neck Pain (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 32
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 29
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 27
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 14
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10
Headache (Nervous system disorders) | 32
Dysgeusia (Nervous system disorders) | 27
Neuropathy Peripheral (Nervous system disorders) | 20
Dizziness (Nervous system disorders) | 14
Peripheral Sensory Neuropathy (Nervous system disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 35
Dehydration (Metabolism and nutrition disorders) | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 6
Hypokalaemia (Metabolism and nutrition disorders) | 6
Insomnia (Psychiatric disorders) | 22
Depression (Psychiatric disorders) | 21
Anxiety (Psychiatric disorders) | 12
Neutropenia (Blood and lymphatic system disorders) | 24
Anaemia (Blood and lymphatic system disorders) | 21
Sinusitis (Infections and infestations) | 15
Upper Respiratory Tract Infection (Infections and infestations) | 13
Urinary Tract Infection (Infections and infestations) | 12
Hypertension (Vascular disorders) | 29
Hot Flush (Vascular disorders) | 6
Weight Decreased (Investigations) | 12
Aspartate Aminotransferase Increased (Investigations) | 8
Alanine Aminotransferase Increased (Investigations) | 7
Neutrophil Count Decreased (Investigations) | 7
Proteinuria (Renal and urinary disorders) | 14
Lacrimation Increased (Eye disorders) | 7

LIMITATIONS AND CAVEATS:
The primary endpoint TTP was changed to overall survival (OS) due to issues regarding tumor assessment data based on RECIST and poor response from investigators to related queries that developed after the planned interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.